CLINICAL TRIAL: NCT00795782
Title: Prophylactic Central Lymph Node Dissection in Papillary Thyroid Microcarcinoma: A Prospective Randomized Controlled Trial
Brief Title: Prophylactic Central Lymph Node Dissection in Papillary Thyroid Microcarcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-09-048
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2011-07

CONDITIONS: Thyroid Cancer
Keywords: Papillary thyroid carcinoma; Lymph node dissection; Lymph node metastasis; Prophylactic node dissection; Central lymph node metastasis
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary; Lymphatic Metastasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- UniCND (Experimental): Limited/ipsilateral central lymph node dissection
  Interventions: Procedure: Prophylactic central lymph node dissection
- BiCND (Active Comparator): Comprehensive/bilateral central lymph node dissection
  Interventions: Procedure: Prophylactic central lymph node dissection
- NoCND (No Intervention): No central lymph node dissection

INTERVENTIONS:
Procedure: Prophylactic central lymph node dissection — prophylactic ipsilateral versus bilateral central lymph node dissection
  Arms: BiCND; UniCND

SUMMARY:
The purpose of this study is to determine whether the prophylactic ipsilateral central lymph node dissection is equally effective in the management of papillary thyroid microcarcinoma(PTMC) to the bilateral central lymph node dissection.

DETAILED DESCRIPTION:
The extent, the advantage and disadvantage of prophylactic central lymph node dissection was not fully established up to now in papillary thyroid microcarcinoma.

Prophylactic bilateral central lymph node dissection can give a important clinical information about the status of lymph nodes, and possibly guide a further adjuvant treatment. However, it causes high postoperative morbidity, including hypocalcemia and hoarseness. In this respect, some advocate no central lymph node dissection in prophylactic settings.

Thus, we aimed to prove the efficacy of prophylactic ipsilateral central lymph node dissection in thyroid papillary microcarcinoma, compared to the bilateral dissection and no dissection.

Type of Study design: Prospective randomized, controlled double-blinded (to subjects and observers) study.

Group I: Limited/ipsilateral central lymph node dissection (UniCND) Group II: Comprehensive/bilateral central lymph node dissection (BiCND) Group III: No central lymph node dissection (NoCND)

Outcomes: vocal cord palsy, hypocalcemia, locoregional recurrence, distant metastasis

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 70
* Sonographically node-negative cytology confirmed thyroid papillary carcinoma
* Tumor size less than 1 cm in sonography
* Tumor confined to the one lobe of the thyroid gland
* One who provides the informed consent

Exclusion Criteria:

* History of radiation treatment to head and neck area
* History of other malignancy except thyroid cancer
* Poor performance status (ECOG 3-4)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Recurrence (Thyroglobulin level, antiTG level, results of follow-up imaging tools) | 3 year after initial treatment

SECONDARY OUTCOMES:
Postoperative complications(hypocalcemia, hoarseness) | up to 3 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Han-Sin Jeong, MD, PhD, Principal Investigator — Samsung Medical Center, Department of Otorhinolaryngology-Head and Neck Surgery
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Son YI, Jeong HS, Baek CH, Chung MK, Ryu J, Chung JH, So YK, Jang JY, Choi J. Extent of prophylactic lymph node dissection in the central neck area of the patients with papillary thyroid carcinoma: comparison of limited versus comprehensive lymph node dissection in a 2-year safety study. Ann Surg Oncol. 2008 Jul;15(7):2020-6. doi: 10.1245/s10434-008-9928-8. Epub 2008 May 6. PMID 18459004